CLINICAL TRIAL: NCT06200779
Title: Susceptibility-guided Vs. Empirical First-line Bismuth Quadruple Therapy of H. Pylori Infection: a National Prospective Multicentric Randomized Controlled Trial.
Brief Title: Tailored Vs. Empirical Helicobacter Pylori Infection Treatment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Manuel Coelho da Rocha (Other)
Responsible Party: Sponsor-Investigator, Manuel Coelho da Rocha, Principal Investigator, Unilabs Portugal
Organization: Unilabs Portugal (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clinical Study Protocol 1
Record Dates: First submitted 2023-12-12; First posted 2024-01-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Antibiotic resistance; Eradication treatment; Molecular pathology
MeSH Terms: interventions — Mutation; Amoxicillin; Clarithromycin; WW Domain-Containing Oxidoreductase; Levofloxacin

STUDY DESIGN:
Intervention Model Description: Intervention group: Patients will receive a prescription for oriented H. pylori eradication treatment according to the following rules: a) clarithromycin-sensitive strain (independently of levofloxacin resistance test result) - PPI, amoxicillin 1 g and clarithromycin 500 mg, twice daily, for 10 days; b) clarithromycin-resistant and levofloxacin-sensitive strain - PPI, amoxicillin 1g and levofloxacin 250 mg, twice daily, for 10 days; c) clarithromycin-resistant and levofloxacin-resistant strain - bismuth quadruple therapy (Pylera®) for 10 days.
  Control Group: Patients will receive a prescription for empirically H. pylori eradication treatment with bismuth quadruple therapy (Pylera®) for 10 days.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Patients randomized to the Intervention group will receive a prescription for oriented H. pylori eradication treatment according to the following rules: a) clarithromycin-sensitive strain (independently of levofloxacin resistance test result) - PPI, amoxicillin 1 g and clarithromycin 500 mg, twice daily, for 10 days; b) clarithromycin-resistant and levofloxacin-sensitive strain - PPI, amoxicillin 1g and levofloxacin 250 mg, twice daily, for 10 days; c) clarithromycin-resistant and levofloxacin-resistant strain - bismuth quadruple therapy (Pylera®) for 10 days. At least 4 weeks after stopping antibiotics (and at least 2 weeks after stopping PPIs), an eradication control test will be carried out using a respiratory test (urea breath test) or endoscopic biopsies (if clinical indication for that).
  Interventions: Diagnostic Test: Clarithromycin (mutations in the 23S rRNA gene, A2134G, A2142G and A2142C mutations) and levofloxacin resistance (mutations in the gyrA gene) PCR test; Drug: PPI, amoxicillin 1 g and clarithromycin 500 mg, twice daily, for 10 days; Drug: PPI, amoxicillin 1g and levofloxacin 250 mg, twice daily, for 10 days; Drug: Bismuth quadruple therapy (Pylera®) for 10 days
- Control group (Active Comparator): Patients randomized to the Control group will receive a prescription for empirically H. pylori eradication treatment with bismuth quadruple therapy (Pylera®) for 10 days. At least 4 weeks after stopping antibiotics (and at least 2 weeks after stopping PPIs), an eradication control test will be carried out using a respiratory test (urea breath test) or endoscopic biopsies (if clinical indication for that).
  Interventions: Drug: Empirically H. pylori eradication treatment with bismuth quadruple therapy (Pylera®)

INTERVENTIONS:
Diagnostic Test: Clarithromycin (mutations in the 23S rRNA gene, A2134G, A2142G and A2142C mutations) and levofloxacin resistance (mutations in the gyrA gene) PCR test — Described in "Arms" section
  Arms: Intervention group
Drug: Empirically H. pylori eradication treatment with bismuth quadruple therapy (Pylera®) — Described in "Arms" section
  Arms: Control group
Drug: PPI, amoxicillin 1 g and clarithromycin 500 mg, twice daily, for 10 days — Administered to patients randomized to Intervention group and with H. pylori clarithromycin-sensitive strain
  Arms: Intervention group
Drug: PPI, amoxicillin 1g and levofloxacin 250 mg, twice daily, for 10 days — Administered to patients randomized to Intervention group and with H. pylori clarithromycin-resistant and levofloxacin-sensitive strain
  Arms: Intervention group
Drug: Bismuth quadruple therapy (Pylera®) for 10 days — Administered to patients randomized to Intervention group and with H. pylori clarithromycin-resistant and levofloxacin-resistant strain
  Arms: Intervention group

SUMMARY:
Helicobacter pylori (Hp) is a gram-negative bacterium that colonizes human gastric mucosa and is associated with chronic gastritis that can progress to severe complications such as peptic ulcer disease, gastric adenocarcinoma and gastric mucosa-associated lymphoid tissue lymphoma. More than half of the world's population is infected with H. pylori and Portugal is one of the countries with the highest Hp burden. All of infected patients should be treated, however, H. pylori treatment is challenged by the continuously rising antibiotic resistance which has reached alarming levels worldwide. For this reason, it is now well accepted that tailoring treatment of H. pylori infection based on systematic antimicrobial susceptibility testing is useful to avoid the increase of antibiotic resistance.

Our aims are to determine prospectively the efficacy and safety of first-line H. pylori eradication treatment based on resistance profile (determined by molecular methods) vs. empirical bismuth quadruple therapy, to evaluate the accuracy of H. pylori detection by polymerase chain reaction (PCR) (vs. histopathological examination) and to estimate the prevalence of H. pylori infection and H. pylori resistance to clarithromycin and levofloxacin in Portugal.

This prospective study will be the first national study to investigate the benefits of tailored H. pylori eradication treatment. The investigators expect that this project will be able to demonstrate the non-inferiority of susceptibility-guided treatment comparing with empirical therapy, and our results may change H. pylori treatment recommendations by systematically applying antibiotic susceptibility testing before prescribing eradication therapy.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized, controlled interventional trial in two arms: intervention group and control group.

Eligible patients will receive oral and written information and will be enrolled after giving written informed consent.

In all patients complete gastroscopy with white light will be performed and endoscopic findings will be recorded. For each patient, gastric body and antral biopsies will be collected. All gastric samples will be tested for H. pylori infection by histopathological examination and PCR. All H. pylori positive samples will be tested for clarithromycin (mutations in the 23S rRNA gene, A2134G, A2142G and A2142C mutations) and levofloxacin resistance (mutations in the gyrA gene) by PCR.

All H. pylori positive patients will be randomized in two groups:

INTERVENTION GROUP: Patients randomized to the Intervention group will receive a prescription for oriented H. pylori eradication treatment according to the following rules: a) clarithromycin-sensitive strain (independently of levofloxacin resistance test result) - PPI, amoxicillin 1 g and clarithromycin 500 mg, twice daily, for 10 days; b) clarithromycin-resistant and levofloxacin-sensitive strain - PPI, amoxicillin 1g and levofloxacin 250 mg, twice daily, for 10 days; c) clarithromycin-resistant and levofloxacin-resistant strain - bismuth quadruple therapy (Pylera®) for 10 days. At least 4 weeks after stopping antibiotics (and at least 2 weeks after stopping PPIs), an eradication control test will be carried out using a respiratory test (urea breath test) or endoscopic biopsies (if clinical indication for that).

CONTROL GROUP: Patients randomized to the Control group will receive a prescription for empirically H. pylori eradication treatment with bismuth quadruple therapy (Pylera®) for 10 days. At least 4 weeks after stopping antibiotics (and at least 2 weeks after stopping PPIs), an eradication control test will be carried out using a respiratory test (urea breath test) or endoscopic biopsies (if clinical indication for that).

All patients that complete eradication treatment regimen will be evaluated 2 to 4 weeks after performing the eradication control (urea breath test) in a clinical consultation. Eventual adverse effects will be recorded. A negative breath test will define the success of the treatment, while a positive test will define treatment failure. The latter will be managed according to H. pylori infection guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 years old scheduled for upper GI endoscopy with indication for gastric biopsies (clinical or endoscopic findings)

Exclusion Criteria:

* 1st phase (clinical): patients who had received antimicrobial therapy 1 month prior to endoscopy; patients who had received proton pump inhibitor (PPI) therapy 2 weeks prior to endoscopy; patients who had ever received H. pylori eradication therapy (despite its efficacy); history of previous gastrectomy; non-Portuguese nationality; pregnant or breastfeeding women; women of childbearing age without effective contraception; suspected or documented allergy to amoxicillin; serious comorbidities (ASA 3 or more); ongoing medication with anticoagulants
* 2nd phase (endoscopic): upper GI tract neoplasia; hemorrhagic gastritis; upper GI tract varices
* 3rd phase (pathological): H. pylori negative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of successful H. pylori eradication treatment in intervention group vs. control group. | 12 months
  This comparation will allow the investigators to show the non-inferiority of susceptibility-guided treatment comparing with empirical therapy

SECONDARY OUTCOMES:
Percentage of H. pylori detection in gastric samples by PCR vs. histopathological examination. | 12 months
  All gastric samples will be tested for H. pylori infection by histopathological examination and PCR. This comparation will allow the investigators to analyze tha diagnostica accuracy of PCR vs. histopathological examination
Estimate the prevalence of H. pylori infection in Portugal. | 12 months
Estimate the prevalence of H. pylori resistance to clarithromycin and levofloxacin in Portugal. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unilabs Portugal, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting in May 2025